CLINICAL TRIAL: NCT00504049
Title: Wavelet Analysis of Surface EMG in Cerebral Palsy
Brief Title: Wavelet Analysis of Electromyography (EMG) in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Richard T. Lauer, Shriners Hospitals for Children
Other Study IDs: 1R03NS048875-01A2 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Electromyography; Wavelet Analysis
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Several methods exist to evaluate motor function in the child with cerebral palsy and are used to assess the outcome of a clinical intervention. However, these scales are not directed towards measuring the changes in muscle activity patterns that can result from the intervention. For example, there are classification scales aimed at measuring motor function and functional abilities, and indices of gait function. These scores, while providing a way to quantify function and mechanics, do not directly measure muscle activation characteristics. Therefore, these tests may be insensitive to how the intervention has directly affected muscle function, which is usually the focus of the intervention (i.e. botulinum toxin, functional electrical stimulation, dorsal rhizotomy). Muscle biopsies and motor evoked potentials can provide information about the muscle activation characteristics, however, they are invasive and there are concerns about using these techniques on the pediatric population and/or the practicality of clinical implementation, especially since they do not provide insight into how the muscle behaves during a functional task. One method that can be used to provide insight into muscle activity in a non-invasive and clinically meaningful manner is the use of surface electromyography (sEMG). Surface EMG is typically a routine part of clinical assessment and the evaluation of motor impairment in CP. However, the analysis of the data has been limited in most cases to examination of signal amplitude or differences in muscle onset and offset timing.

The long-term goal of this research is to develop an analysis method for sEMG that can be used during functional tasks for treatment planning, diagnostic, assessment purposes in CP. This is to be accomplished through the use of the continuous wavelet transform (CWT). By developing an assessment method based on muscle activity, it is believed that a clinically viable measurement tool can be devised that will provide a level of insight into the effects of an intervention on muscle pathophysiology that is not currently available. The first step in progressing towards this long-term goal is to determine the variability and range of expected time-frequency patterns that can be expressed in a given population (i.e., cerebral palsy) during the execution of a meaningful task (gait), and relate the time-frequency information back to more standard assessments

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of spastic diplegic CP
* Must be ambulatory without the use of orthotics
* Between a GMFCS Level I and Level III
* Between the ages of 7 and 13 years
* Cleared by an orthopedic surgeon for risk of hip subluxation or dislocation and cannot have significant scoliosis (curvature > 40 degrees)
* Seizure-free or seizure controlled
* Has visuoperceptual skills and cognitive/communication skills sufficient to follow multiple step commands and to attend to tasks associated with data collection
* Must be greater than 1 year post-surgery to the lower extremities
* Must be greater then 6 months botulinum toxin injection
* Passive range of motion in lower extremity joints must be greater than 10 degrees of flexion contracture at the hips as measured by the Thomas Test, at least 20 degrees of hip abduction bilaterally, less than 5 degrees of knee flexion contracture, popliteal angle less than 45 degrees, and at least 0 degrees of ankle dorsiflexion with the knee extended while the foot is in varus

Exclusion Criteria:

* Children who do not meet the inclusion criteria will not be considered for the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with spastic, diplegic cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-03; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lauer, PhD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Philadelphia, Pennsylvania, United States